CLINICAL TRIAL: NCT02046785
Title: Comparison of CVP Values , ΔPP and Echocardiographic at Different Angles Headwaters Before and After Volume Challenge
Brief Title: Hemodynamic Measurements at Different Inclinations of the Head
Acronym: HMDIH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Rosangela de Oliveira Felice, nursing specialist, Federal University of Uberlandia
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: Hemodinamica
Record Dates: First submitted 2013-07-11; First posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Hypovolemic Shock
Keywords: Fluid administration; Cardiac output; Right atrial pressure; Resuscitation
MeSH Terms: conditions — Shock | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 0.9% saline solution (Other): comparing values obtained before and after administration of 500 ml of 0.9% saline
  Interventions: Other: 0.9% saline solution

INTERVENTIONS:
Other: 0.9% saline solution — comparing values obtained before and after administration of 500 ml of 0.9% salin
  Other Names: Solution of 0.9% NaCl in distilled water

SUMMARY:
The purpose of this study is to determine whether hemodynamic measures vary in angles bedside before and after volume challenge.

DETAILED DESCRIPTION:
* Check if values of central venous pressure (CVP), pulse pressure variation (Δpp), heart rate (HR), mean arterial pressure ((PAM) vary in different angles headboards
* Compare values of CVP, Δpp, HR and MAP as predictors of blood volume after supply of 500 ml of 0.9% saline solution.

ELIGIBILITY:
Inclusion Criteria:

* Being in circulatory shock and have at least one of the following criteria to identify loss of tissue perfusion: systolic blood pressure <90 mmHg or need for vasoactive drugs, urine output below 0.5 ml / kg / h.
* Being under sedation, assessed by the scale of Richmond agitation and sedation (RASS) -5, mechanically ventilated in volume control mode with tidal volume between 8 to 12 ml/kg, PEEP to 8 cm H2O.
* Tue signing the informed consent by legal guardian.

Exclusion Criteria:

* Presence cardiac arrhythmias.
* Presence of abdominal or thoracic trauma.
* Contraindication for passive elevation of the members.
* Hypoxia significant PaO2/FiO2 < or equal 100.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Different Backrest position's effect on CVP, CO and ∆PP measures | Data collection was performed at admission or within 10 days of hospitalization between September 2013 and February 2014.

CONTACTS AND LOCATIONS:
Overall Officials: Rosangela O Felice, expert, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Intensive Care Unit, Clinical Hospital, Federal University of Uberlandia, Uberlândia, Minas Gerais, Brazil